CLINICAL TRIAL: NCT02064270
Title: Prospective Randomized, Controlled Study to Assess Prevention of Incision Healing Complications in Patients Undergoing Total Knee or Hip Arthroplasty, Treated With Either Negative Pressure Wound Therapy or Standard Dressings.
Brief Title: Study to Compare Negative Pressure Wound Therapy or Standard Dressings After Orthopedic Surgery
Acronym: PICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, James Stannard, Medical Director, Missouri Orthopaedic Institute; Chairman, Department of Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1208434
Record Dates: First submitted 2014-02-06; First posted 2014-02-17 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Wound of Knee; Wound of Hip
Keywords: incision care; Total Hip Arthroplasty; Total Knee Arthroplasty; Knee surgery; Hip surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): Single-Use Negative Pressure Wound Therapy (NPWT)
  Interventions: Device: Single-Use Negative Pressure Wound Therapy
- Standard dressings (Active Comparator): Standard postsurgical dressings
  Interventions: Device: Standard postsurgical dressings

INTERVENTIONS:
Device: Single-Use Negative Pressure Wound Therapy — Application of PICO Single-Use Negative Pressure Wound Therapy
  Other Names: NPWT; PICO
  Arms: Negative Pressure Wound Therapy
Device: Standard postsurgical dressings — Use of Standard postsurgical dressings
  Arms: Standard dressings

SUMMARY:
The aim of this study is to assess the prevention of incision healing complications in patients undergoing Total Knee Arthroscopy (TKA) and Total Hip Arthroscopy (THA) treated with either Single-Use Incisional NPWT (Negative Pressure Wound Therapy), or standard of care dressings.

DETAILED DESCRIPTION:
Most surgical wounds heal by primary intention, meaning the wound edges are brought together, or approximated, by some sort of mechanical means (sutures, staples, paper tape, surgical glue or adhesive strips) to heal with minimal scar formation. National clinical guidelines recommend that incisions are covered with a postsurgical cover dressing, for up to a period of 48 hours, to help control postoperative bleeding, absorb exudate, provide mechanical protection, help to reduce edema and provide protection from exogenous sources. Multiple patient comorbidities, environmental factors and the type and length of surgery may elevate certain groups of patients into a higher level of risk of developing a post-surgical complication: calling for a higher degree of vigilance and postsurgical intervention. Surgical complications include; wound dehiscence, infection (deep or superficial), hematomas, seromas, tissue necrosis and delayed incision healing. Complication rates can range from 19% in patients requiring open reduction and internal fixation (ORIF) of tibial plateau, pilon and calcaneus fractures up to 50% in high energy trauma wounds. These complications can have a high degree of morbidity for the patient and further sequelae may result in additional surgical procedures or revisions, a lower functional status for the patient, an increased in length of hospital stay (LOS) and a higher cost for the healthcare provider.

Traditional NPWT has been shown to be an effective adjunct therapy in the treatment of acute and chronic wounds, but the emergence of incisional NPWT (iNPWT) and supporting evidence is growing momentum. In vitro studies have shown that iNPWT may help to improve the stimulation of blood flow, help manage exudate, help to reduce edema, provide a mechanical and "splinting" effect on the incision and provide mechanical protection from the environment. Its impact on the prevention or reduction of post-surgical incision complications is still in its infancy, but recent studies have been encouraging and have demonstrated a statistically significant reduction in infection and dehiscence in patients considered as high-risk following severe skeletal trauma.

The aim of this study is to assess the prevention of incision healing complications in patients undergoing TKA and THA treated with either Single-Use Incisional NPWT compared to standard of care dressings.

ELIGIBILITY:
Inclusion Criteria:

1. - Patient ≥18 years old
2. - Male or non-pregnant females
3. - Patient is scheduled to have a surgical procedure for Total Knee Arthroplasty or Total Hip Arthroplasty (Primary or Revision Procedure)
4. - The patient is able to understand the trial and is willing to consent to the trial

Exclusion Criteria:

1. - Patients who in the opinion of the investigator may not complete the study for any reason
2. - Patients with a known history of poor compliance with medical treatment
3. - Patients who have participated in this trial previously and who were withdrawn
4. - Patients with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing)
5. - Patients not capable of obtaining a standardized digital picture at day 7 (1 week from surgery), and submitting it to the site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2014-03; Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Stannard, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Started | 263 | 263
Completed | 201 | 231
Not Completed | 62 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings | Total
Number analyzed (Participants) | 201 | 231 | 432
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [33 to 86] | 60.5 [35 to 82] | 60.6 [33 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 137 | 263
  Male | 75 | 94 | 169
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 201 | 231 | 432

OUTCOME MEASURES:

1. Primary Outcome: Incision Appearance Based on VAS (Incision Healing Assessment Form)
Description: Visual Analog Pain Scale (VAS): PICO Study Incision Healing Assessment Form. Used to represent the assessment of incision healing based on in-person visual appearance, or appearance based on standard digital photograph. This number is reported as a total score on a 0-100 scale, with 0 being poor incision healing and 100 being excellent incision healing.
Time Frame: 35 days (+/- 14 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Number analyzed (Participants) | 201 | 231
units on a scale | 83.4 (13.3) | 83.5 (12.2)

2. Secondary Outcome: Drainage Amount
Description: Incision Drainage:
  1. None
  2. Slight (barely noticed)
  3. Moderate (significant amount, but did not have to change dressing)
  4. Extensive (had to change dressing)
Time Frame: 35 days (+/- 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Number analyzed (Participants) | 194 | 223
Participants
  None | 178 | 211
  Slight (barely noticed) | 9 | 9
  Moderate (significant amount, but did not have to | 4 | 2
  Extensive (had to change dressing) | 3 | 1

3. Secondary Outcome: User-friendliness for Patient
Description: User-Friendliness of PICO device:
  1. Easy to use (no difficulties, no instruction needed)
  2. Slightly difficult (needed instruction)
  3. Minor difficulties (but able to use effectively)
  4. Difficult (not able to use effectively)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy
Number analyzed (Participants) | 131
Participants
  Easy to use | 113
  Slightly difficult | 11
  Minor difficulties | 7
  Difficult | 0

4. Secondary Outcome: Number of Participants With Complications
Description: Complications experienced by the subject within the study period time-frame will be recorded.
Time Frame: 35 days (+/- 14 days)
Measure: Number; unit: participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Number analyzed (Participants) | 201 | 231
participants | 27 | 41

5. Secondary Outcome: Return to the Operating Room
Description: Information regarding the subject returning to the operating room within the research study time-frame will be recorded.
Time Frame: 35 days (+/- 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Number analyzed (Participants) | 193 | 222
Participants
  Return to OR | 193 | 4
  No Return to OR | 0 | 218

6. Secondary Outcome: Need for Antibiotics
Description: The need for additional antibiotics will be recorded.
Time Frame: 35 days (+/- 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
Number analyzed (Participants) | 193 | 223
Participants
  Need for additional antibiotics | 25 | 30
  No need for additional antibiotics | 168 | 193

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Negative Pressure Wound Therapy | Standard Dressings
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/231
Serious Adverse Events (participants affected / at risk) | 5/201 | 6/231
Other Adverse Events (participants affected / at risk) | 3/201 | 5/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Wound Therapy (N=201) | Standard Dressings (N=231)
Deep Infection Requiring Additional Surgery (Surgical and medical procedures) | 5 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Negative Pressure Wound Therapy (N=201) | Standard Dressings (N=231)
Superficial Infection (Infections and infestations) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02064270/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02064270/Prot_SAP_001.pdf